CLINICAL TRIAL: NCT04012736
Title: Physical Fitness in Celiac Disease Patients - the Effect of a Gluten Free Diet
Status: Terminated | Type: Observational
Why Stopped: Inability to recruit and perform study visits due to COVID19 pandemic
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, eyal zifman, Head of Pediatric Gastroenterology Service, Meir Medical Center
Other Study IDs: MMC059-19CTIL
Record Dates: First submitted 2019-06-24; First posted 2019-07-09 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Celiac Disease in Children
Keywords: gluten free diet; fitness; pediatric

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Celiac disease: Celiac disease subjects enrolled after diagnosis and before gluten free diet initiation
- Control: Healthy controls with no chronic condition

SUMMARY:
Evaluating the effect of Celiac disease (CD) and gluten free diet (GFD) on physical fitness parameters among CD subjects. The CD subjects will be compared to healthy controls.

DETAILED DESCRIPTION:
This is a prospective observational cohort study. The study would take place at Meir Medical Center (Kfar-Saba, Israel), a secondary-level academic hospital. The investigators will enroll 50 newly diagnosed CD subjects. The diagnosis will be in accordance with the European Society for Gastroenterology Hepatology and Nutrition guidelines for the diagnosis of CD from 2012 (6). The investigators will also enroll 50 control subjects. The control subjects are children visiting the pediatric gastroenterology clinic. Before enrollment the investigators will rule out chronic conditions involving the gastrointestinal tract including CD.

All subjects will be enrolled after providing an informed consent and signing the consent form.

The investigators will obtain the following measurements and evaluations at and 6 months after enrollment:

1. Anthropometric measurements: Height, weight, body mass index (BMI) and total body fat will be evaluated using a TANITA scale. The z-score for each parameter will be recorded.
2. A Godin leisure-time exercise questionnaire (7) will be filled by the subjects and their parents
3. Evaluation of physical fitness by the Eurofit fitness testing (8). This series of physical fitness tests was developed to evaluate speed, stamina and strength in school-aged children.

   1. Flamingo balance test
   2. Seat and reach test
   3. Standing broad jump test
   4. Handgrip test
   5. Sit-ups test
   6. Bent arm hang test
   7. Twenty meter endurance shuttle run test
   8. Wingate anaerobic fitness test
4. Bone speed of sound test will be performed by a bone sonometer - a non-invasive ultrasound based measurement of bone density.
5. CD subjects will be evaluated for adherence to GFD via questioning by a pediatric gastroenterologist and a clinical dietitian and by serum tissue transglutaminase immunoglobulin A (IgA) level (or serum deamidated gliadin peptide immunoglobulin G level in IgA deficient subjects). This is part of the normal follow-up of CD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 4-18y visiting the pediatric gastroenterology clinic
2. Signing a consent form

Exclusion Criteria:

1. Family history of cardiovascular diseases or sudden death before age 50y
2. Chronic condition limiting the ability to perform the physical fitness tests (e.g. juvenile idiopathic arthritis)
3. Failure to complete the measurements and evaluations by 2 months from the date of the visit at the clinic

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The investigators will enroll 50 newly diagnosed CD subjects. The diagnosis will be in accordance with the European Society for Gastroenterology Hepatology and Nutrition guidelines for the diagnosis of CD from 2012. The investigators will also enroll 50 control subjects. The control subjects are children visiting the pediatric gastroenterology clinic. Before enrollment the investigators will rule out chronic conditions involving the gastrointestinal tract including CD.
  All subjects will be enrolled after providing an informed consent and signing the consent form.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Flamingo balance test | 6 months
  Flamingo balance test recorded in times in 60sec (n).
Sit and reach test | 6 months
  Sit and reach test recorded in cm.
Standing broad jump test | 6 months
  Standing broad jump test recorded in cm.
Handgrip test | 6 months
  Handgrip test recorded kg.
Sit-ups test | 6 months
  Sit-ups test is recorded in times in 30sec (n).
Bent arm hang test | 6 months
  Bent arm hang test recorded in sec.
Twenty meter endurance shuttle run test | 6 months
  Twenty meter endurance shuttle run test recorded in times (n).

SECONDARY OUTCOMES:
Weight | 6 months
  Weight in kilograms. Measured with an electronic scale (model 500KL, Health o meter, McCook, IL, USA). Range 0-220kg, rounded to the nearest 0.1kg.
Height | 6 months
  Height in centimeters. Measured with a wall-mounted stadiometer (model 240, Seca, Hamburg, Germany). Range 0-240cm, rounded to the nearest 0.1cm.
Body mass index | 6 months
  Weight and height will be combined to report BMI in kg/m^2
Total body fat | 6 months
  Total body fat in percents. Measured with a body composition scale (model MC-780U, Tanita, Arlington Heights, IL, USA).
Bone speed of sound | 6 months
  Bone speed of sound in m/s. Measured with a bone sonometer (Sunlight Omnisense, Somerset, NJ, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Zifman, MD, Principal Investigator — Meur Medical Center, Kfar-Saba, Israel
Locations (1):
- Meir Medical Center, Kfar Saba, Israel